CLINICAL TRIAL: NCT06781333
Title: A Pilot Study to Assess the Effect of Adding 1 Infusion of Human Mesenchymal Stem Cells (hMSC) to the Treatment of Patients Suffering Agitation/Aggression or Other Behavioral Abnormalities From Alzheimer's Disease.
Brief Title: Human Mesenchymal Stem Cells (hMSC) in Behavioral Problems Due to Alzheimer's Disease.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bernard (Barry) Baumel (Other)
Responsible Party: Sponsor-Investigator, Bernard (Barry) Baumel, Associate Professor of Neurology, University of Miami
Organization: University of Miami (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20240984
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-03

CONDITIONS: Alzheimer Disease; Agitation in Dementia
Keywords: aggression; behavior; agitation
MeSH Terms: conditions — Alzheimer Disease; Aberrant Motor Behavior in Dementia; Aggression; Behavior; Psychomotor Agitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- hMSC group (Experimental): Participants in this group will receive one infusion of hMSC. Total participation is up to 12 weeks.
  Interventions: Biological: hMSC

INTERVENTIONS:
Biological: hMSC — Participants will come in person to receive one intravenous infusion of approximately 25 million cells up to 20 minutes.

SUMMARY:
The purpose of this research study is to test if adding one infusion of mesenchymal stem cells to the current treatment with antipsychotic medication may help control behavioral problems in people with a diagnosis of moderate to severe Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Adults 55-90 years at the time of signing consent
* A diagnosis of probable Alzheimer disease (AD), defined by the National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria
* Previous computed tomography or magnetic resonance imaging scan of the brain with findings consistent with a diagnosis of Alzheimer disease
* A diagnosis of behavioral symptoms that include any of the following: delusions, hallucinations, agitation/aggression, depression/dysphoria, anxiety, elation/euphoria, apathy/indifference, disinhibition, irritability/lability, aberrant motor behavior, sleep and nighttime behavior disorders and appetite and eating disorders
* Onset of behavioral symptoms at least 4 weeks prior to screening.
* Treatment with antipsychotic medication for at least 4 weeks prior to the hMSC infusion.
* Patients unable to consent should have a Legally Authorized Representative or Proxy to provide consent on their behalf.
* Have a family member or friend (study partner) who has frequent and sufficient contact with the patient and able to answer questions about the participant's behavior.

Exclusion Criteria:

* Dementia other than AD
* Patient with severe depression. Patient with controlled depression is allowed to participate.
* Recent history of substance abuse
* History of bleeding disorders, HIV, Hepatitis C Virus or Hepatitis B Virus
* Recent history (within 3 years) of malignancies, except for treated basal cell, squamous carcinoma or melanoma in situ, prostate in situ, cervical carcinoma in situ.
* Uncontrolled medical conditions (hypertension, diabetes, unstable angina or Myocardial Infarction within 1 year prior to screening)
* History of bleeding disorder
* Currently receiving (or received within four weeks of screening) experimental agents for the treatment of Alzheimer's Disease or enrolled in clinical trials in the prior 3 months.
* Be a transplant recipient or in any other active medical condition than in the opinion of the investigator may compromise the safety or compliance of the patient or preclude successful completion of the study
* Be premenopausal

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Neuropsychiatric Inventory | Up to 12 weeks.
  Score ranges from 0-12, higher scores indicate a worse psychiatric outcome

SECONDARY OUTCOMES:
Change in antipsychotic medications dosage | Baseline to 12 weeks
  Will be measured in milligrams
Change in number of antipsychotic medications | Baseline to 12 weeks
  Will be measured in number of antipsychotic medications

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Baumel, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Department of Neurology, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No